CLINICAL TRIAL: NCT03328871
Title: The Combination Therapy of Fractional Laser and Platelet-Rich Plasma Injection Compared With Nanofat Grafting and Platelet-Rich Plasma Synergy in Treating Striae Gravidarum.
Brief Title: The Combination Therapy of Fractional Laser and PRP Compared With Nanofat Grafting and PRP Synergy in Treating Striae Gravidarum.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First Affiliated Hospital of Jinan University (Other)
Collaborators: Science and Technology Program of Guangzhou (Unknown)
Responsible Party: Principal Investigator, Li-Ling Xiao, Associate Chief of Department of Plastic Surgery,The First Affiliated Hospital of Jinan University, Guangzhou, First Affiliated Hospital of Jinan University
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LXiao FirstJinanU
Record Dates: First submitted 2017-09-26; First posted 2017-11-01 (Actual); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Treatments of Striae Gravidarum
Keywords: Striae Gravidarum; Fractional Laser; Platelet-Rich Plasma (PRP); Nanofat Graft; Combination Therapy
MeSH Terms: conditions — Striae Distensae | interventions — Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fractional CO2 Laser and PRP injection (Experimental): One of the striae gravidarum areas will be treated by fractional laser once every three months for 2 times combined with PRP injection once a month for 6 times.
  Interventions: Device: Fractional CO2 Laser; Procedure: Platelet-rich plasma (PRP) Injection
- Nanofat grafting and PRP injection (Experimental): Another area will be treated by nanofat grafting once every three months for 2 times and PRP therapy once a month for 6 times.
  Interventions: Procedure: Nanofat grafting; Procedure: Platelet-rich plasma (PRP) Injection

INTERVENTIONS:
Device: Fractional CO2 Laser — Fractional Carbon Dioxide Laser will be treated once every three months for 2 times.
  Arms: Fractional CO2 Laser and PRP injection
Procedure: Nanofat grafting — Nanofat grafting will be applied once every three months for 2 times.
  Arms: Nanofat grafting and PRP injection
Procedure: Platelet-rich plasma (PRP) Injection — PRP Injection will be applied once a month for 6 times.

SUMMARY:
Nowadays, multiple treatment modalities have been applied clinically to treat striae gravidarum, such as laser therapy, microdermabrasion, platelet-rich plasma injection(PRP), etc. To some extent, these treatments can improve striae gravidarum. In this clinical trial, the investigators are going to treat striae gravidarum by using two different kinds of combination therapies. One is fractional laser and PRP injection synergy, and the other one is treated by nanofat grafting with PRP injection.

DETAILED DESCRIPTION:
The investigators will pick out two areas of most severe striae gravidarum on a participant's abdomen. One of the areas will be treated by fractional laser once every three months for 2 times combined with PRP injection once a month for 6 times. Another area will be treated by nanofat grafting once every three months for 2 times and PRP therapy once a month for 6 times. The participants were asked to come back 1、3、6、9 months after treatment for further follow-up.

Before and after the treatment, the striae gravidarum will be assessed subjectively by satisfaction assessment, dermatoscope and ultrasound, and objectively by immunohistochemical analysis.

ELIGIBILITY:
Inclusion Criteria:

* The striae gravidarum was appeared within 3 years
* Age ≤ 35 years old
* Not in lactation
* Not pregnancy within one year

Exclusion Criteria:

* Skin allergy
* Skin inflammation or wound
* Platelet dysfunction syndrome
* Take anticoagulant drugs
* Acute or chronic infection
* Chronic liver disease
* Photodermatosis
* Active vitiligo, psoriasis, systemic lupus erythematosus
* Other clinical trial

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Immunohistochemical analysis | Baseline and 15 months.
  The tissue extracted will be taken for immunohistochemical analysis to observe the change of epidermal and dermal thickness, and the distribution and amount of elastic fiber and collagen fiber,etc.

SECONDARY OUTCOMES:
Dermatoscope | Baseline and at 3,6,9,12,15 months after the treatments.
  The striae gravidarum will be assessed by dermatoscope to observe the pigmentation condition of striae after the application of laser or nanofat grafting with PRP injection.
Ultrasound | Baseline and at 3,6,9,12,15 months after the treatments.
  The striae gravidarum will be assessed by ultrasound in order to observe the change of dermal thickness of striae after the application of laser or nanofat grafting with PRP injection.

OTHER OUTCOMES:
Satisfaction assessments | After every sessions of treatments, and at 6,9,12,15 months.
  The participants, investigators and physicians will fill in a satisfaction assessment about any complication during the treatments.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Jinan University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cervelli V, Nicoli F, Spallone D, Verardi S, Sorge R, Nicoli M, Balzani A. Treatment of traumatic scars using fat grafts mixed with platelet-rich plasma, and resurfacing of skin with the 1540 nm nonablative laser. Clin Exp Dermatol. 2012 Jan;37(1):55-61. doi: 10.1111/j.1365-2230.2011.04199.x. PMID 22182435
- [Background] Kamakura T, Kataoka J, Maeda K, Teramachi H, Mihara H, Miyata K, Ooi K, Sasaki N, Kobayashi M, Ito K. Platelet-Rich Plasma with Basic Fibroblast Growth Factor for Treatment of Wrinkles and Depressed Areas of the Skin. Plast Reconstr Surg. 2015 Nov;136(5):931-939. doi: 10.1097/PRS.0000000000001705. PMID 26171752
- [Background] Mehryan P, Zartab H, Rajabi A, Pazhoohi N, Firooz A. Assessment of efficacy of platelet-rich plasma (PRP) on infraorbital dark circles and crow's feet wrinkles. J Cosmet Dermatol. 2014 Mar;13(1):72-8. doi: 10.1111/jocd.12072. PMID 24641609
- [Background] Kim IS, Park KY, Kim BJ, Kim MN, Kim CW, Kim SE. Efficacy of intradermal radiofrequency combined with autologous platelet-rich plasma in striae distensae: a pilot study. Int J Dermatol. 2012 Oct;51(10):1253-8. doi: 10.1111/j.1365-4632.2012.05530.x. PMID 22994672
- [Background] Tonnard P, Verpaele A, Peeters G, Hamdi M, Cornelissen M, Declercq H. Nanofat grafting: basic research and clinical applications. Plast Reconstr Surg. 2013 Oct;132(4):1017-1026. doi: 10.1097/PRS.0b013e31829fe1b0. PMID 23783059
- See also: Treatment of traumatic scars using fat grafts mixed with platelet-rich plasma, and resurfacing of skin with the 1540 nm nonablative laser. — http://pubmed.cn/22182435
- See also: Platelet-Rich Plasma with Basic Fibroblast Growth Factor for Treatment of Wrinkles and Depressed Areas of the Skin. — http://pubmed.cn/26171752
- See also: Assessment of efficacy of platelet-rich plasma (PRP) on infraorbital dark circles and crow's feet wrinkles. — http://pubmed.cn/24641609
- See also: Efficacy of intradermal radiofrequency combined with autologous platelet-rich plasma in striae distensae: a pilot study. — http://pubmed.cn/22994672
- See also: Nanofat grafting: basic research and clinical applications. — http://pubmed.cn/23783059

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-21): https://cdn.clinicaltrials.gov/large-docs/71/NCT03328871/Prot_SAP_000.pdf